CLINICAL TRIAL: NCT06888778
Title: Efficacy of Deep-coil Based Repetitive Transcranial Magnetic Stimulation in the Treatment of Parkinson's Disease With Freezing of Gait and Its Neural Regulation Mechanism Study of Resting-state Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, Guangli Ren, Associate Director of Neurology, Ningbo Medical Center Lihuili Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2022PJ280
Record Dates: First submitted 2025-02-17; First posted 2025-03-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Parkinson disease; Freezing of Gait; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimulation group (Experimental): participants receive repetitive transcranial magnetic stimulation (rTMS)
  Interventions: Other: repetitive transcranial magnetic stimulation (rTMS)
- Non-stimulation group (Placebo Comparator): participants receive Non-stimulation:The side of the double cone coil is placed against the scalp, and the target of the coil is stimulated in the direction of air.
  Interventions: Other: Non-stimulation

INTERVENTIONS:
Other: repetitive transcranial magnetic stimulation (rTMS) — rTMS is a non-invasive brain stimulation technique that stimulates specific brain areas through repeated magnetic pulses to treat depression, anxiety and other mental illnesses, and to study brain function.
  Arms: stimulation group
Other: Non-stimulation — participants receive Non-stimulation:The side of the double cone coil is placed against the scalp, and the target of the coil is stimulated in the direction of air.
  Arms: Non-stimulation group

SUMMARY:
The protocol for repetitive transcranial magnetic stimulation (rTMS) in treating Parkinson's disease (PD) with freezing of gait (FOG) has not yet established an internationally unified standard, and the heterogeneity of treatment parameters is often the main factor leading to significant differences in efficacy. Based on descriptive analyses and existing data from studies with relatively small sample sizes, the current research primarily focuses on unilateral stimulation targets, without exploring the effectiveness of stimulating the bilateral primary motor centers for lower limbs (M1-LL). Moreover, most studies use figure-of-eight coils or circular coils, while deep-coil stimulation may be more effective for M1-LL. There is still a lack of research employing arterial spin labeling (ASL) imaging to explore the neural mechanisms of resting-state cerebral blood flow (CBF) regulation associated with rTMS treatment for FOG.

Therefore, this research project will focus on improving the above - mentioned issues. The high - frequency stimulation of bilateral M1 - LL using a deep - coil (double - cone coil) will be selected. The sample size will be further expanded to evaluate the efficacy of rTMS in treating freezing of gait (FOG). Combined with the three - dimensional arterial spin labeling (3D - ASL) imaging technique, the changes in resting - state cerebral blood flow (CBF) before and after treatment will be analyzed to explore the possible neural mechanisms of rTMS in treating FOG.

DETAILED DESCRIPTION:
Magstim rapid 2 transcranial magnetic stimulation instrument was used with double-cone coils, and the stimulation target was bilateral M1-LL. The total stimulation time of each target was 10 minutes, once a day, 5 times a week (5 consecutive working days), and the treatment was continuous for 2 weeks, a total of 10 times.

Stimulus parameter setting:

* True stimulus group: 100% Rest Motor Threshold (RMT), 10Hz, each stimulus lasted 10 seconds, 55 seconds apart, a total of 10 strings. Once a day, each side of the lower extremity region of the primary motor cortex received a total of 1000 pulses.
* In the pseudo-stimulation group, the side of the double-cone coil was placed against the scalp, and the bull 's-eye of the coil was stimulated towards the air. Other treatment parameters were the same as those of true stimulation group.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the clinical diagnostic criteria for Parkinson's disease established by the Movement Disorder Society (MDS) in 2015.
* Aged between 45 and 70 years old, regardless of gender.
* Regularly taking anti - Parkinson's disease medications for a long time (≥3 years), accompanied by freezing of gait, and with poor efficacy of medications;
* A score of ≥24 on the Mini - Mental State Examination (MMSE).
* Signing the informed consent form and being willing to actively cooperate with the treatment.

Exclusion Criteria:

* Freezing of gait caused by parkinsonism and parkinson plus syndromes.
* Having a history of central nervous system diseases such as cerebral infarction, cerebral hemorrhage, leukoencephalopathy, and migraine.
* Having been diagnosed with epilepsy or having had epileptic seizures.
* Having undergone craniocerebral surgery, having cerebral aneurysms or arteriovenous malformations, having metal implants in the skull, or having had a cardiac pacemaker implanted.
* Having a history of other mental illnesses or a family history of mental illnesses, such as schizophrenia, bipolar disorder, autism, mental retardation, depression, etc.
* Having received rTMS treatment.
* Severe PD (H&Y grade ≥ 4).
* Severe organ dysfunction or severe physical diseases.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Within 24 hours before treatment, within 24 hours after treatment, and 1 month after treatment
  In this study, Unified Parkinson's Disease Rating Scale(UPDRS) score was used as an assessment tool for PD patients. Four subscales, UPDRS II (0-52 scores), UPDRS III (0-56 scores), UPDRS V (0-5 grades), and UPDRS VI (0-11 grades), were used to assess the condition. The higher the score or grade, the sicker the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Medical Center Li Huili Hospital, Ningbo, China, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rascol O, Brooks DJ, Korczyn AD, De Deyn PP, Clarke CE, Lang AE. A five-year study of the incidence of dyskinesia in patients with early Parkinson's disease who were treated with ropinirole or levodopa. N Engl J Med. 2000 May 18;342(20):1484-91. doi: 10.1056/NEJM200005183422004. PMID 10816186